CLINICAL TRIAL: NCT00416104
Title: Postcesarean Section Pain: Possible Demographic and Medical Predictors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Other Study IDs: zimmerctil
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2006-12-27 (Estimated); Status verified 2006-07

CONDITIONS: Pain; Cesarean Section
Keywords: analgesia
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The aim of this retrospective study is to find out if one or more of the following parameters has an impact on postcesarean section pain:age,ethnic origin, parity,body habitus, smoking, breastfeeding, education,newborn in intensive care unit, primary/repeated operation,elective/emergency operation,junior/senior surgeon,type of anesthesia during operation.

DETAILED DESCRIPTION:
The medical records of 600 consecutive women with a cesarean section will be reviewed.We will analyse the correlations between postcesarean section pain levels,analgesic consumption and; age,ethnic origin, parity,body habitus, smoking, breastfeeding, education,newborn in intensive care unit, primary/repeated operation,elective/emergency operation,junior/senior surgeon,type of anesthesia during operation.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing a cesarean section

Exclusion Criteria:

* Medical or psychological conditions not enabling reliable patients pain assessment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2006-12; Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: etan z zimmer, MD, Principal Investigator — director of obstetrics rambam medical center
Locations (1):
- Rambam Medical Center, Haifa, Israel